CLINICAL TRIAL: NCT03395873
Title: A Phase I Study of Avelumab in Combination With Decitabine as First Line Treatment of Patients With AML, Who Are Unfit for Intensive Chemotherapy
Brief Title: Avelumab With Decitabine as First Line for AML Treatment of Patients With AML, Who Are Unfit for Intensive Chemotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recent FDA approval of a new drug for the same patient population
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Hong Zheng, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSCI 17-033
Record Dates: First submitted 2017-12-28; First posted 2018-01-10 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — avelumab; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): * Decitabine 20mg/m2 IV day 1-5, every 28 days
  * Avelumab 10mg/kg IV, day 1, every 14 days
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — * Decitabine 20mg/m2 IV day 1-5, every 28 days
  * Avelumab 10mg/kg IV, day 1, every 14 days
  Other Names: Decitabine

SUMMARY:
The goal of this study is to test the safety of combination treatment with Avelumab and Decitabine in newly diagnosed AML patients who are unfit for intensive induction chemotherapy.

DETAILED DESCRIPTION:
This is a single arm, open label phase I study with expansion to evaluate safety and tolerability of Avelumab in combination with Decitabine in patients with untreated AML, who are unfit for intensive chemotherapy. Decitabine will be given 20mg/m2 IV day 1-5, every 28 days. Avelumab will be given at 10mg/kg IV (initial dose) day 1, every 14 days. Using a standard 3x3 statistical design, protocol defined Dose Limiting Toxicities (DLT) will be assessed. In expansion stage, we will perform an expansion cohort of 9 additional patients using the Maximum Tolerated Dose (MTD) established in the Phase I portion.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically or histologically confirmed diagnosis of AML (except M3 acute promyelocytic leukemia) according to WHO classification.
2. Previously untreated AML except for hydroxyurea.
3. Age ≥18 years. Because no dosing or adverse event data are currently available on the use of avelumab in combination with decitabine in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric trials.
4. Performance status (ECOG) of 0-2 (see Appendix A).
5. Not considered candidates for intensive remission induction chemotherapy at time of enrollment based on EITHER:

   * 75 years of age OR <75 years of age with at least 1 of the following: Poor performance status (ECOG) score of 2.

   Clinically significant heart or lung comorbidities, as reflected by at least 1 of:

   Left ventricular ejection fraction (LVEF) ≤50%. Lung diffusing capacity for carbon monoxide (DLCO) ≤65% of expected. Forced expiratory volume in 1 second (FEV1) ≤65% of expected. Chronic stable angina or congestive heart failure controlled with medication. Liver transaminases >3 × upper limit of normal (ULN). Other contraindication(s) to anthracycline therapy. Other comorbidity the investigator judges incompatible with intensive remission induction chemotherapy. The enrollee declines intensive remission induction chemotherapy.
6. Creatinine clearance as estimated by the Cockcroft-Gault (C-G) or other medically acceptable formulas ≥30 mL/min.vii. Cytogenetic features justify hypo-methylating agents as induction treatment.
7. Life expectancy > 12 weeks (3months).
8. Patients may not have received prior azacytidine or decitabine for MDS that has transformed to AML.
9. Hydroxyurea would be permitted for control of elevated WBC prior to treatment and can be continued for the first 4 weeks of therapy.
10. Women of childbearing potential (not surgically sterile or one year postmenopausal) must have a negative result for a serum pregnancy test before study drug administration on cycle 1 day 1 (within 3 days). Women of childbearing potential (not surgically sterile or one year postmenopausal) must use a highly effective method of contraception and must agree to continue use of this method for the duration of the study and for 30 days after discontinuation of study drug. Acceptable methods of contraception include abstinence, barrier method with spermicide, intrauterine device (IUD) known to have a failure rate of less than 1% per year, or steroidal contraceptive (oral, transdermal, implanted, or injected) in conjunction with a barrier method.
11. The patient, if a man, is surgically sterile or, if capable of producing offspring, is currently using an approved method of birth control and agrees to continued use of this method for the duration of the study (and for 30 days after taking the last dose of study drug because of the possible effects on spermatogenesis). Acceptable methods of contraception include abstinence, female partner's use of steroidal contraceptive (oral, implanted or injected) in conjunction with a barrier method, female partner's use of an IUD known to have a failure rate of less than 1% per year, or if female partner is surgically sterile or one year post- menopausal. In addition, male patients may not donate sperm for the duration of the study and for 30 days after taking study drug.
12. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Patients who are receiving any other investigational agents.
3. Patients should be excluded if they have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
4. Patients with known CNS involvement will be excluded because of poor prognosis and concerns regarding progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
5. History of severe hypersensitivity reaction to any monoclonal antibody.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant women are excluded from this study because avelumab is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with avelumab, breastfeeding should be discontinued if the mother is treated with avelumab.
8. Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) might be enrolled if the viral load by PCR is undetectable with/without active treatment and absolute lymphocyte count >= 350/ul.

   Patients with a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection might be enrolled if the viral load by PCR is undetectable with/without active treatment.
9. Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as SLE, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjögren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
10. Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event).
11. Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if <10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
12. Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study.
13. Prior organ transplantation including allogenic stem-cell transplantation.
14. Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines.
15. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
16. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
17. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Safety of Avelumab in combination with decitabine in AML. | 28 days
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
The complete remission (CR+CRi) rate. | 4months
  Response will be determined by bone marrow aspiration.
The overall survival (OS). | 2 years
  Percentage of participates who are alive at 2 years from enrollment will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zheng, MD, Principal Investigator — Penn State Cancer Institute
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States